CLINICAL TRIAL: NCT06459518
Title: Effectiveness of Bowen Technique vs Muscle Energy Technique in Mechanical Neck Pain Among Desktop Users.
Brief Title: Effectiveness of Bowen Technique vs Muscle Energy Technique in Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01106
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain; Musculoskeletal Manipulation
Keywords: Bowen Therapy; Mechanical Neck Pain; Muscle Energy Technique
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen Therapy along with Conventional Therapy (Experimental): Group A will receive Bowen Therapy along with Conventional Therapy
  Interventions: Other: Bowen Therapy along with conventional therapy
- Muscle Energy Technique along with conventional Therapy (Active Comparator): Group B will receive Muscle Energy Technique along with Conventional Therapy
  Interventions: Other: Muscle Energy Technique with Conventional Therapy

INTERVENTIONS:
Other: Bowen Therapy along with conventional therapy — Bowen Technique Group Assignment: Participants will be assigned to undergo targeted Bowen Technique therapy sessions.
  Session Details: The therapy sessions will include:
  * Gentle, rolling-type maneuvers
  * Specific placements of fingers and thumbs
  * Focus on muscles, tendons, and ligaments associated with neck pain Therapeutic Pauses: There will be intentional pauses between sets of moves to allow the body time to respond to the therapeutic stimulation.
  Conventional Therapy: Hot pack, TENS, Passive Stretching 2 times a week for 4 weeks
  Arms: Bowen Therapy along with Conventional Therapy
Other: Muscle Energy Technique with Conventional Therapy — MET Session Structure: Participants will engage in Muscle Energy Technique (MET) sessions that focus on:
  * Isometric muscle contractions, where muscles are contracted without changing length.
  * Therapist-guided, controlled contractions against specific resistance.
  * Relaxation Periods: Each contraction session will be followed by a period of relaxation to allow muscles to recover and respond to the therapy.
  conventional therapy: Hot pack, TENS, Passive Stretching 2times a week for 4 weeks.
  Arms: Muscle Energy Technique along with conventional Therapy

SUMMARY:
Mechanical neck pain, also known as non-specific neck pain, is a prevalent ailment that results from problems with spine and surrounding tissue function. Trauma, degenerative changes, strained muscles, and bad posture are among the causes. The range of symptoms includes headaches, stiffness, and mild to severe pain. The goal of treatment is to strengthen the muscles and improve posture. The diagnosis is clinical. The Bowen Technique is a type of gentle bodywork therapy that promotes relaxation and overall rebalancing by using specific movements to activate the autonomic nerve system. It is sought for the improvement of general well-being, pain alleviation, and stress reduction. Patients undergoing manual treatment will be asked to actively contract their muscles against regulated resistance using the Muscle Energy Technique (MET). It addresses problems including joint limitations and attempts to return muscles and joints to their normal functions.

DETAILED DESCRIPTION:
The research, will last for ten months at the Limit Institute of Health Sciences in Sahiwal, is a randomized controlled trial. With 10 participants in each group using a non-probability convenient sampling procedure, the sample size includes 10% attrition. Computer users between the ages of 18 and 35 who work five to seven hours a day meet the inclusion criteria, but recent musculoskeletal injuries and a history of head or spine trauma are the exclusion criteria. One instrument used to collect data is the Neck Disability Index (NDI). There are two established study groups: Group B will receive Muscle Energy Technique (MET) and traditional physiotherapy, while Group A will receive Bowen therapy and conventional physiotherapy. Blinding will be used, and the study will adhere to a recruitment, enrollment, and randomization procedure. SPSS version 23 will be used to analyze the data, and descriptive statistics, change over temporal analysis as well as tests of group comparison. The purpose of the study is to evaluate how the interventions affect people who use computers for extended periods in terms of their functional results and mechanical neck discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Computer users who work 5-7 hours daily.
* Age between 18 to 35 will be included.
* Both genders

Exclusion Criteria:

* Any recent musculoskeletal injury of upper limb or spine.
* History of any trauma of spine or head

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain level | 4th week
  The Numeric Pain Rating Scale (NPRS) is a straightforward tool used to measure pain intensity in adults, including those suffering from chronic pain associated with rheumatic conditions. It features an 11-point scale, where '0' indicates no pain and '10' signifies the most extreme pain possible, described as "pain as bad as you can imagine" or "the worst pain imaginable."
Functional Disability | 4th week
  A self-reported questionnaire called the Neck Disability Index (NDI) is used to gauge how neck pain affects a person's ability to function and go about their everyday life. It is divided into eleven sections that address different tasks such as sleeping, work, reading, lifting, and personal care. In each category, respondents rate the level of difficulty they encounter; scores are added together to produce a percentage that indicates the degree of disability. When conducting clinical assessments, the NDI is a useful instrument that helps medical practitioners determine the degree of functional limits and provide personalized interventions for patients with neck discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Wajeeha Saeed, DPT, Principal Investigator — Riphah International University
Locations (1):
- Maryam Polyclinic Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masaracchio M, Kirker K, States R, Hanney WJ, Liu X, Kolber M. Thoracic spine manipulation for the management of mechanical neck pain: A systematic review and meta-analysis. PLoS One. 2019 Feb 13;14(2):e0211877. doi: 10.1371/journal.pone.0211877. eCollection 2019. PMID 30759118
- [Background] Verhagen AP. Physiotherapy management of neck pain. J Physiother. 2021 Jan;67(1):5-11. doi: 10.1016/j.jphys.2020.12.005. Epub 2020 Dec 24. No abstract available. PMID 33358545
- [Background] Joshi S, Balthillaya G, Neelapala YVR. Thoracic Posture and Mobility in Mechanical Neck Pain Population: A Review of the Literature. Asian Spine J. 2019 Jun 3;13(5):849-860. doi: 10.31616/asj.2018.0302. Print 2019 Oct. PMID 31154701
- [Background] Al-Khazali HM, Kroll LS, Ashina H, Melo-Carrillo A, Burstein R, Amin FM, Ashina S. Neck pain and headache: Pathophysiology, treatments and future directions. Musculoskelet Sci Pract. 2023 Aug;66:102804. doi: 10.1016/j.msksp.2023.102804. Epub 2023 Jun 16. PMID 37394323
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Bonilla-Barba L, Florencio LL, Rodriguez-Jimenez J, Falla D, Fernandez-de-Las-Penas C, Ortega-Santiago R. Women with mechanical neck pain exhibit increased activation of their superficial neck extensors when performing the cranio-cervical flexion test. Musculoskelet Sci Pract. 2020 Oct;49:102222. doi: 10.1016/j.msksp.2020.102222. Epub 2020 Jul 11. PMID 32861371